CLINICAL TRIAL: NCT00036504
Title: Efficacy and Safety of Twice-Daily Insulin Lispro Low Mixture Compared to a Once-Daily Long Acting Insulin Comparator in Patients New to Insulin Therapy Who Were Inadequately Controlled on Oral Agents
Brief Title: Efficacy and Safety of Twice-Daily Insulin Lispro Low Mixture Compared to a Once-Daily Long Acting Insulin Comparator in Patients Who Have Been Using One or More Oral Antihyperglycemic Agents Without Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4050; F3Z-MC-IOND
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus, insulin deficiency, hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia

INTERVENTIONS:
Drug: Insulin Lispro low mixture

SUMMARY:
The purposes of this study are to determine: 1. If patients taking insulin lispro LM with metformin will have better overall control of their blood sugar than patients taking a long acting insulin comparator with metformin. 2. If there is a difference in the way the two treatments affect blood sugar control before and after meals and at night. 3. If there is a difference in the insulin dose required with the two treatments. 4. If there is a difference in the numbers of times patients experience low blood sugar with the two treatments. 5. If there is a difference in the effect on patients's body weight.

DETAILED DESCRIPTION:
The aim of the present study is to compare two treatments - LM twice daily plus metformin two or three times daily versus a long acting insulin comparator once daily plus metformin two or three times daily - in patients with type 2 diabetes who are currently using a regimen of one or more oral antihyperglycemic agents.

The primary objective of this study is to demonstrate that, in patients with type 2 diabetes who are new to insulin, hemoglobin A1c at endpoint will be lower after treatment with insulin lispro LM twice daily plus metformin than after treatment with a long acting insulin comparator once daily plus metformin.

This will be a multicenter, randomized, open-label, crossover study comparing twice-daily insulin lispro LM plus two- or three-times-daily metformin to a once-daily long acting insulin comparator plus two- or three-times-daily metformin in patients with type 2 diabetes who were receiving one or more oral antihyperglycemic agents without insulin prior to the study.

Following an 8 (+-2) week lead-in period consisting of treatment with NPH once daily at bedtime plus metformin two or three times daily, approximately 100 eligible patients will be randomized to one of two sequence groups, so that there are approximately 50 patients in each group. One group will receive 4 months of insulin lispro LM administered immediately before the morning and evening meals plus metformin two or three times daily followed by 4 months of a once-daily long acting insulin comparator at bedtime plus metformin two or three times daily. The other group will receive the reverse sequence.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes.
* At least 30 years old and less than 80 years old.
* Using oral agents without insulin for 30 days prior ot study.
* Willing to start insulin injections using a pen device.
* Keep a patient diary.

Exclusion Criteria:

* Undergoing therapy for cancers.
* History of renal transplant or receiving renal dialysis.
* Have participated in an interventional medical, surgical, or pharmaceutical study (a study in which a medical or surgical treatment was given) within 30 days prior to entry into the study.
* Women who are breastfeeding.
* Have been treated with a drug within the last 30 days that has not received regulatory approval.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-08; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - La Jolla, California
  - Walnut Creek, California
  - New Britain, Connecticut
  - Longwood, Florida
  - Atlanta, Georgia
  - Fayetteville, Georgia
  - Boise, Idaho
  - Springfield, Illinois
  - Mount Laurel, New Jersey
  - New Brunswick, New Jersey
  - Syracuse, New York
  - Chattanooga, Tennessee
  - Dallas, Texas

REFERENCES:
- [Result] Malone JK, Kerr LF, Campaigne BN, Sachson RA, Holcombe JH; Lispro Mixture-Glargine Study Group. Combined therapy with insulin lispro Mix 75/25 plus metformin or insulin glargine plus metformin: a 16-week, randomized, open-label, crossover study in patients with type 2 diabetes beginning insulin therapy. Clin Ther. 2004 Dec;26(12):2034-44. doi: 10.1016/j.clinthera.2004.12.015. PMID 15823767
- [Result] Hirsch IB, Yuan H, Campaigne BN, Tan MH. Impact of prandial plus basal vs basal insulin on glycemic variability in type 2 diabetic patients. Endocr Pract. 2009 May-Jun;15(4):343-8. doi: 10.4158/EP08308.ORR. PMID 19454394
- [Result] Chan JY, Leyk M, Frier BM, Tan MH. Relationship between HbA1c and hypoglycaemia in patients with type 2 diabetes treated with different insulin regimens in combination with metformin. Diabetes Metab Res Rev. 2009 Mar;25(3):224-31. doi: 10.1002/dmrr.929. PMID 19156705
- [Result] Shrom D, Sarwat S, Ilag L, Bloomgarden ZT. Does A1c consistently reflect mean plasma glucose? J Diabetes. 2010 Jun;2(2):92-6. doi: 10.1111/j.1753-0407.2010.00066.x. Epub 2010 Jan 22. PMID 20923490
- [Result] Sarwat S, Ilag LL, Carey MA, Shrom DS, Heine RJ. The relationship between self-monitored blood glucose values and glycated haemoglobin in insulin-treated patients with Type 2 diabetes. Diabet Med. 2010 May;27(5):589-92. doi: 10.1111/j.1464-5491.2010.02955.x. PMID 20536957